CLINICAL TRIAL: NCT02726464
Title: Testing the Characteristics of Platelet Rich Plasma in Sports Medicine
Acronym: PRiSM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: LightIntegra Technology (Industry)
Responsible Party: Sponsor
Other Study IDs: H16-00328
Record Dates: First submitted 2016-03-29; First posted 2016-04-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Musculoskeletal Pain; Osteoarthritis
Keywords: Platelet-rich Plasma; Cell-Derived Microparticles; Pain Management; Blood Platelets; Therapeutics; Inflammation; ThromboLUX; Dynamic Light Scattering
MeSH Terms: conditions — Musculoskeletal Pain; Osteoarthritis; Agnosia; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study that evaluates the characteristics of Platelet Rich Plasma used in the therapy and treatment of musculoskeletal injuries and degenerative joint diseases.

A sample of the PRP will be tested for platelet and microparticle content using dynamic light scattering to determine if there is a relationship between the composition and the treatment outcome.

DETAILED DESCRIPTION:
An observational study that evaluates the characteristics of Platelet Rich Plasma used in the therapy and treatment of musculoskeletal and degenerative joint conditions.

Patients enrolled in this study have already been assessed by the Principal Investigator and are schedule to receive treatment with Platelet Rich Plasma. Prior to the treatment patients will be asked to consent in the study where the composition of the PRP is to be evaluated. Consenting patients that meet inclusion/exclusion criteria will complete a pain score self-assessment prior to treatment.

An autologous preparation of PRP sample will be made from the subject's whole blood. The subject will receive the PRP treatment and an excess portion of the PRP preparation will be tested for composition and the relative concentration of the constituents.

The sample of the PRP will be tested using Dynamic Light Scattering (ThromboLUX System) to measure the constituents in PRP preparations prior to injection. PRP and whole blood (at physician's discretion) will be analyzed on a hematology analyzer.

The testing work-flow does not alter the subject's standard of care. The physician will be blinded to the analytical results during the enrolment, treatment and patient follow-up phase of the study. Analytical results are not used in patient management decisions.

Patient's response to the PRP treatment will be assessed at 3 and 6 weeks post injection. At these times, the clinical outcome of the treatment will be measured using a patient self -assessment (post-treatment pain scores).

This study will test the hypothesis that PRP characteristics, such as platelet and microparticle content and composition can be predictive clinical outcome for PRP treatments.

The clinical outcome will be evaluated by patient pre- and post-pain score assessment. This study aims to review clinical outcomes and compare these results against ThromboLUX and other test results. If the predictive value of platelet composition testing can be demonstrated, additional studies may be considered.

ELIGIBILITY:
Inclusion Criteria:

* Are willing and able to give informed consent for participation in the study
* Have a diagnosed injury/condition requiring PRP injection: patients with acute or chronic musculoskeletal injury, tendinopathy, or mild to moderate osteoarthritis of the knee
* Are otherwise healthy
* Agree to pre-treatment fasting (4 hours prior to treatment)
* Agree to disclose medications taken in the last 2 weeks
* Able (in the Investigators opinion) and willing to comply with all study requirements
* Able to attend an on-site visit or provide information on your current status electronically, 3 and 6 weeks following the PRP injection
* Have not previously received a PRP injection for your current injury

Exclusion Criteria:

* Unable to provide informed consent
* Have any blood borne disease, currently or in the past
* Have a systemic inflammatory disease, skin or joint infection, bleeding disorders, or compromised immune function
* Have a known platelet abnormality or hematological disorder
* Are not able or willing to share with the study team any medications taken in the last two weeks.
* Taking anti-inflammatory medications or medications that interfere with clotting
* Are female and are pregnant or breast feeding
* Have inadequate venous access for drawing blood
* Have any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the patients ability to participate in the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adults have been selected to receive platelet-rich plasma (PRP) injections as a treatment for musculoskeletal or degenerative joint conditions
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Change in pre- and post- pain score at 3 and 6 weeks | Up to 6 weeks after injection
  The primary objective of the study is to test the hypothesis that the constituents in platelet-rich plasma (PRP) preparations, such as platelet and microparticle content and composition, can be correlated to the clinical outcome for PRP treatments.
The impact of microparticle content on pain scores | Up to 6 weeks after injection
  The study will ascertain the capability of ThromboLUX microparticle assay results to correlate with the clinical outcome for PRP treatments when evaluated by patient pre- and post-pain score assessment.

SECONDARY OUTCOMES:
Correlation of platelet count to ThromboLUX results | Up to 6 weeks after injection
  Evaluation of PRP platelet count to clinical outcome and ThromboLUX data outputs
The use of dynamic light scattering (ThromboLUX) as a patient screening tool | Up to 6 weeks after injection
  To verify the performance of the ThromboLUX instrument in a clinical setting by reviewing size and composition of constituents in PRP

CONTACTS AND LOCATIONS:
Overall Officials: Don McKenzie, MD, PhD, LLD, Principal Investigator — University of British Columbia; Jennifer Leung, MSc, Study Director — LightIntegra Technology Inc
Locations (1):
- Allan McGavin Sports Medicine Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: Patient Brochure — http://www.lightintegra.com/prism-study